CLINICAL TRIAL: NCT00266630
Title: Efficacy and Safety of Olanzapine in the Extended Treatment for Manic or Mixed Episode of Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9637; F1D-JE-BMEX (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Results first posted 2010-06-29 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Manic or Mixed Episode Associated With Bipolar I Disorder
MeSH Terms: conditions — Mania | interventions — Olanzapine; Lithium; Valproic Acid; Carbamazepine

ARMS (2):
- Olanzapine Monotherapy (Experimental): Olanzapine extension for Study BMAC patients who completed Visit 8.
  Patients received olanzapine 5-20 mg for 18 weeks.
  Interventions: Drug: olanzapine
- Olanzapine + Mood Stabilizer (Experimental): Olanzapine extension for Study BMAC patients who discontinued at Visit 4 or 5.
  Patients received an initial dose of olanzapine 10 mg for 1 week and subsequent doses of olanzapine 5-20 mg for 17 weeks.
  Patients received one (1) mood stabilizer (lithium, valproate or carbamazepine) for 18 weeks.
  Interventions: Drug: olanzapine; Drug: lithium; Drug: valproate; Drug: carbamazepine

INTERVENTIONS:
Drug: olanzapine — oral, daily
  Other Names: LY170053; Zyprexa
Drug: lithium — Dose adjusted according to local package insert
  Arms: Olanzapine + Mood Stabilizer
Drug: valproate — Dose adjusted according to local package insert
  Arms: Olanzapine + Mood Stabilizer
Drug: carbamazepine — Dose adjusted according to local package insert
  Arms: Olanzapine + Mood Stabilizer

SUMMARY:
The efficacy and safety of the extended treatment to patients with most recent episode manic or mixed who completed previous double blind study (F1D-JE-BMAC [Study BMAC]) will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in and completed Study BMAC (NCT00129220), or those who discontinued Study BMAC at Visit 4 or Visit 5 due to lack of efficacy and for whom the Young Mania Rating Scale (YMRS) total score at the time of discontinuation was not lower than that at baseline of Study BMAC
* Are diagnosed as "294.4x Bipolar I Disorder, Most Recent Episode Manic" or "296.6x Bipolar I Disorder, Most Recent Episode Mixed," as determined by the Mini-International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* Have a diagnosis of diabetes mellitus
* Significant protocol deviation in Study BMAC
* The actual date of the final visit of Study BMAC is 4 days or more later than the scheduled date of first visit in Study BMEX

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- Japan (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okinawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine Monotherapy: Olanzapine extension for Study BMAC patients who completed Visit 8. Patients received olanapine 5-20 mg for 18 weeks.
Period: Overall Study
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Started | 100 | 39
Completed | 58 | 11
Not Completed | 42 | 28
Not completed — Adverse Event | 8 | 6
Not completed — Lack of Efficacy | 1 | 4
Not completed — Entry Criteria not met | 1 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 10 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 19 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer | Total
Number analyzed (Participants) | 100 | 39 | 139
Age Continuous [Mean (Standard Deviation); unit: years] | 41.8 (11.7) | 43.2 (11.1) | 42.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 21 | 80
  Male | 41 | 18 | 59
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 100 | 39 | 139
Region of Enrollment [Number; unit: participants]
  Japan | 100 | 39 | 139
Current Episode - Mixed or Manic [Number; unit: participants] — Description of the bipolar episode the participant experienced when enrolling into the study.
  participants
    Manic | 88 | 39 | 127
    Mixed | 12 | 0 | 12
Current Episode - Psychotic or Nonpsychotic [Number; unit: participants] — Description of the bipolar episode the participant experienced when enrolling into the study.
  participants
    Psychotic | 13 | 9 | 22
    Nonpsychotic | 87 | 30 | 117
Rapid Cyclers [Number; unit: participants] — A rapid cycler is defined as a person who experiences four or more mood swings or episodes in a twelve-month period.
  participants
    Rapid Cyclers | 7 | 3 | 10
    Non-Rapid Cyclers | 93 | 36 | 129
Clinical Global Impressions - Bipolar Version, Severity of Illness (CGI-BP) overall [Mean (Standard Deviation); unit: units on a scale] — Measures severity of the patient's overall severity of bipolar symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
  units on a scale | 1.9 (1.0) | 4.7 (0.8) | 2.7 (1.6)
Hamilton Depression Scale - 17 item version (HAMD-17) Total Score [Mean (Standard Deviation); unit: units on a scale] — The 17-item HAMD measures depression severity. Each item was evaluated and scored using a 3-point scale (e.g. absent, mild, marked) or a 5-point scale (e.g. absent, mild, moderate, severe, very severe). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
  units on a scale | 1.8 (3.1) | 4.4 (3.9) | 2.5 (3.5)
Length of Current Episode [Mean (Standard Deviation); unit: days] | 33.5 (23.9) | 35.0 (26.7) | 33.9 (24.6)
Mean Age at Onset of Illness [Mean (Standard Deviation); unit: years] | 31.5 (11.6) | 29.8 (8.4) | 31.0 (10.8)
Young Mania Rating Scale (YMRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
  units on a scale | 5.7 (6.4) | 33.2 (6.6) | 13.4 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint in Young Mania Rating Scale (YMRS) Total Scores - Olanzapine Monotherapy Arm Only
Description: The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60. The primary objective was only interested in the effects in the olanzapine monotherapy arm.
Time Frame: baseline through 18 weeks
Population: The primary objective was only interested in the effects in the olanzapine monotherapy arm, thus the results for the olanzapine + mood stabilizer arm are presented as secondary outcomes. Analyzed were all participants in the olanzapine monotherapy arm who had baseline and post-baseline measurements. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine Monotherapy
Number analyzed (Participants) | 100
units on a scale | -3.0 (5.6)
Statistical Analysis 1: Comparison: Olanzapine Monotherapy; Test type: Superiority or Other; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-4.10 to -1.90]

2. Primary Outcome: Number of Participants With Response of Manic Symptoms - Olanzapine Monotherapy Arm Only
Description: Defined by a 50% or more reduction in YMRS total score from baseline in Study BMAC to endpoint. The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60. The primary objective was only interested in the effects in the olanzapine monotherapy arm.
Time Frame: baseline through 18 weeks
Population: Analyzed were all participants in the olanzapine monotherapy arm who had baseline and post-baseline measurements. Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy
Number analyzed (Participants) | 100
participants | 97

3. Primary Outcome: Number of Participants With Remission of Mania - Olanzapine Monotherapy Arm Only
Description: Remission of Mania was defined as a YMRS total score of less than or equal to 12 at endpoint. The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60. The primary objective was only interested in the effects in the olanzapine monotherapy arm.
Time Frame: baseline through 18 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy
Number analyzed (Participants) | 100
participants | 93

4. Primary Outcome: Number of Participants With Relapse of Manic Symptoms - Olanzapine Monotherapy Arm Only
Description: Patients achieved remission in Study BMAC (defined as YMRS total score <=12 and HAMD-17 total score <=7) and obtained YMRS total score of >=15 at any time during Study BMEX. The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60. The primary objective was only interested in the effects in the olanzapine monotherapy arm.
Time Frame: baseline through 18 weeks
Population: Analyzed were all participants in the olanzapine monotherapy group who were in remission at baseline (end of Study BMAC) with 12 points or less in YMRS total score and 7 points or less in the 17-item Hamilton Depression Rating Scale total score.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy
Number analyzed (Participants) | 79
participants | 3

5. Secondary Outcome: Change From Baseline to Endpoint on the YMRS Total Score - Olanzapine + Mood Stabilizer Only
Description: The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
Time Frame: baseline through 18 weeks
Population: Analyzed were all participants who had baseline and post-baseline measurements. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 39
units on a scale | -19.8 (17.8)
Statistical Analysis 1: Comparison: Olanzapine + Mood Stabilizer; Test type: Superiority or Other; Mean Difference (Final Values) = -19.8, 95% CI 2-sided [-25.58 to -14.06]

6. Secondary Outcome: Clinical Global Impressions - Bipolar Version, Severity of Illness (CGI-BP) Overall, Visit Data
Description: Measures severity of the patient's overall severity of bipolar symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: baseline, Weeks 1, 2, 4, 6, 10, 14, 18
Population: Analyzed were all participants who had baseline and post-baseline measurements. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 100 | 39
units on a scale
  baseline | 1.9 (1.0) | 4.7 (0.8)
  1 week | 1.8 (1.0) | 4.1 (1.2)
  2 weeks | 1.8 (1.0) | 3.7 (1.3)
  4 weeks | 1.7 (1.0) | 3.5 (1.6)
  6 weeks | 1.7 (1.1) | 3.4 (1.7)
  10 weeks | 1.7 (1.1) | 3.0 (1.8)
  14 weeks | 1.8 (1.2) | 3.0 (1.9)
  18 weeks endpoint | 1.7 (1.2) | 2.9 (2.0)

7. Secondary Outcome: Number of Participants Who Experienced Switch to Symptomatic Depression as Measured by the Hamilton Depression Scale - 17 Item Version (HAMD-17)
Description: Incidence of depressive symptoms was defined as a score of equal to or more than 13 points on the HAMD-17. The 17-item HAMD measures depression severity. Each item was evaluated and scored a 3-point scale (e.g. absent, mild, marked) or a 5-point scale (e.g. absent, mild, moderate, severe, very severe). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: baseline through 18 weeks
Population: Analyzed were all participants who had equal to or less than 7 points on the HAMD-17 total score at baseline.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 92 | 30
participants | 4 | 1

8. Secondary Outcome: Number of Participants With Relapse of Depressive Symptoms
Description: Assessed were participants meeting remission criteria for bipolar disorder in Study BMAC and have a HAMD-17 total score greater than or equal to 13 at any time. The 17-item HAMD measures depression severity. Each item was evaluated and scored using a 3-point scale (e.g. absent, mild, marked) or a 5-point scale (e.g. absent, mild, moderate, severe, very severe). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: baseline through 18 weeks
Population: Analyzed were all participants in the olanzapine monotherapy group who had 12 points or less in the YMRS total score and 7 points or less in the HAMD-17 total score at baseline.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy
Number analyzed (Participants) | 79
participants | 4

9. Secondary Outcome: Number of Participants Who Experienced Remission of Bipolar Disorder
Description: Participants who had equal to or less than 12 points in YMRS total score and equal to or less than 7 points in HAMD-17 total score at 18 weeks. YMRS: 11-item scale, measures the severity of manic episodes. 4 items are rated from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total: 0 to 60. The 17-item HAMD measures depression severity. Each item was evaluated and scored using a 3-point scale or a 5-point scale. HAMD-17 total score: 0 (normal) to 52 (severe).
Time Frame: Week 18
Population: Analyzed were all participants who had baseline and post-baseline measurements. Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 100 | 39
participants | 54 | 12

10. Secondary Outcome: Positive and Negative Syndrome Scale Positive Scores - Visit Data
Description: Assesses positive symptoms associated with schizophrenia. 7 items make up the Positive scale. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total Positive Subscale scores range from 7 to 49. For the analysis, the score was converted to 0 to 6 for each item range; hence, the total score ranges from 0 to 42.
Time Frame: baseline, Weeks 1, 2, 4, 6, 10, 14, 18
Population: Analyzed were all participants who had baseline and post-baseline measurements. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 100 | 39
units on a scale
  baseline | 7.7 (1.8) | 12.5 (5.7)
  1 week | 7.5 (1.6) | 10.5 (4.1)
  2 weeks | 7.5 (1.4) | 10.1 (3.9)
  4 weeks | 7.4 (1.4) | 10.1 (5.4)
  6 weeks | 7.3 (1.2) | 10.1 (5.4)
  10 weeks | 7.4 (1.7) | 9.9 (5.4)
  14 weeks | 7.4 (1.7) | 9.9 (5.4)
  18 week endpoint | 7.4 (1.7) | 9.9 (5.4)

11. Secondary Outcome: Number of Participants Who Switched to Syndromic Depression
Description: As defined as a shift from a Manic Episode at baseline to a Major Depressive Episode, at any post baseline visit, based on Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision.
Time Frame: baseline through 18 weeks
Population: Analyzed were all participants who had a manic episode at baseline.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 88 | 39
participants | 8 | 4

12. Secondary Outcome: Maximum Change From Baseline to Endpoint on the Drug Induced Extra-Pyramidal Symptoms Scale (DIEPSS) - Total Score
Description: A scale used to assess the extrapyramidal symptoms attributable to antipsychotics. Consists of 9 items (8 to assess individual symptoms and 1 to assess global severity). Each item is assessed from 0 (none, normal) to 4 (severe). The total points of 8 items are defined as DIEPSS total (0 to 32 points). The items for the assessment of individual symptoms are classified into 4 categories of parkinsonism, akathisia, dystonia and dyskinesia. Parkinsonism is assessed by the total points of items 1 to 5; akathisia, dystonia and dyskinesia are assessed by the points given to the corresponding items.
Time Frame: baseline through 18 weeks
Population: Analyzed were all participants who had baseline and post-baseline measurements. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 100 | 39
units on a scale
  Baseline | 0.35 (1.01) | 0.18 (0.60)
  Maximum Change from baseline to endpoint | 0.05 (1.21) | 0.64 (1.51)

13. Secondary Outcome: Number of Participants With Treatment-Emergent Parkinsonism Based on DIEPSS Scores
Description: DIEPSS assesses the extrapyramidal symptoms attributable to antipsychotics. Consists of 9 items (8 to assess individual symptoms and 1 to assess global severity). Each item is assessed from 0 (none, normal) to 4 (severe). The total points of 8 items are defined as DIEPSS total (0 to 32 points). Parkinsonism is assessed by the total points of items 1 to 5 (total score of 0 to 20). Treatment-emergent parkinsonism was defined as a score of equal or greater than 3 on 1 item, equal or greater than 2 on 2 items, or an increase of equal or greater than 3 from baseline on the parkinsonism total.
Time Frame: baseline through 18 weeks
Population: Included were all participants who did not have an abnormal value at baseline.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 100 | 39
participants | 1 | 3

14. Secondary Outcome: Number of Participants With Treatment-Emergent Akathisia Based on DIEPSS Scores
Description: DIEPSS assesses the extrapyramidal symptoms attributable to antipsychotics. Consists of 9 items (8 to assess individual symptoms and 1 to assess global severity). Each item is assessed from 0 (none, normal) to 4 (severe). The total points of 8 items are defined as DIEPSS total (0 to 32 points). The items are classified into 4 categories of parkinsonism, akathisia, dystonia and dyskinesia. Treatment-emergent akathisia was defined as a score of equal or more than 2 or an increase of equal or more than 2 points from baseline on the akathisia item (total score possible 0 to 4 points).
Time Frame: baseline through 18 weeks
Population: Included were all participants who did not have an abnormal value at baseline.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 98 | 38
participants | 3 | 2

15. Secondary Outcome: Number of Participants With Treatment-Emergent Dystonia Based on DIEPSS Scores
Description: DIEPSS assesses the extrapyramidal symptoms attributable to antipsychotics. Consists of 9 items (8 to assess individual symptoms and 1 to assess global severity). Each item is assessed from 0 (none, normal) to 4 (severe). The total points of 8 items are defined as DIEPSS total (0 to 32 points). The items are classified into 4 categories of parkinsonism, akathisia, dystonia and dyskinesia. Treatment-emergent dystonia was defined as a score equal or more than 2 or an increase of equal or more than 2 points from baseline on the dystonia item (total score possible 0 to 4 points).
Time Frame: baseline through 18 weeks
Population: Included were all participants who did not have an abnormal value at baseline.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 100 | 38
participants | 0 | 1

16. Secondary Outcome: Number of Participants With Treatment-Emergent Dyskenisia Based on DIEPSS Scores
Description: DIEPSS assesses the extrapyramidal symptoms attributable to antipsychotics. Consists of 9 items (8 to assess individual symptoms and 1 to assess global severity). Each item is assessed from 0 (none, normal) to 4 (severe). The total points of 8 items are defined as DIEPSS total (0 to 32 points). The items are classified into 4 categories of parkinsonism, akathisia, dystonia and dyskinesia. Treatment-emergent dyskenisia was defined as a score of equal or more than 2 or an increase of equal to or more than 2 points from baseline on the dyskenisia item (total score possible 0 to 4 points).
Time Frame: baseline through 18 weeks
Population: Included were all participants who did not have an abnormal value at baseline.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 100 | 39
participants | 0 | 0

17. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes in Laboratory Analytes
Description: Triglycerides: high limit equal to or more than 500 milligram/deciliter (mg/dL); Glucose (non-fasting): low limit 2.4975 mmol/liter (L); high limit 13.875 mmol/L; Glucose (fasting): low limit 2.4975 mmol/L; high limit 6.993 mmol/L.
Time Frame: baseline through 18 weeks
Population: Analyzed were all participants without an abnormal value in the direction at baseline (for example, participants with an abnormally low value at baseline who experienced an abnormally low value at any time post baseline were not included, but were included if they experienced an abnormally high value at any time post baseline).
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 100 | 38
participants
  High triglycerides; n=100, n=38 | 5 | 2
  Low glucose (non-fasting); n=64, n=28 | 0 | 0
  High glucose (non-fasting); n=64, n=28 | 0 | 0
  Low glucose (fasting); n=40, n=6 | 0 | 0
  High glucose (fasting); n=40, n=6 | 3 | 0

18. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes in Vital Signs and Weight
Description: Low systolic blood pressure (SBP): <=90 millimeter mercury (mmHg) and decrease of >=20 mmHg; High SBP: >=180 mmHg and increase of >=20 mmHg; Low diastolic blood pressure (DBP): <=50 mmHg and decrease of >=15 mmHg; High DBP: >=105 mmHg and increase of >=15 mmHg; Low pulse: <50 beats per minute (bpm) and decrease of >=15 bpm; High pulse: >120 bpm and an increase of >=15 bpm; Low weight: decrease of >=7%; High weight: increase of >=7%;
Time Frame: baseline through 18 weeks
Population: Analyzed were all study participants.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 100 | 39
participants
  Low systolic blood pressure | 6 | 2
  High systolic blood pressure | 0 | 0
  Low diastolic blood pressure | 4 | 1
  High diastolic blood pressure | 1 | 0
  Low weight | 3 | 1
  High weight | 17 | 10
  Low pulse | 0 | 0
  High pulse | 0 | 0

19. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes in Electrocardiograms - High Fridericia Corrected QT Interval (QTcF)
Description: High QTcF: more than or equal to 450 milliseconds (msec) for males; more than or equal to 470 milliseconds (msec) for females
Time Frame: baseline through 18 weeks
Population: Analyzed were all participants who had baseline and post-baseline measurements and no abnormal values in the direction at baseline (e.g. participants with an abnormally low value for a given parameter at baseline who showed an abnormally low value for the same parameter at a later visit were not included). Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 97 | 39
participants | 0 | 0

20. Secondary Outcome: Number of Participants With Treatment-emergent Abnormal, High, or Low Laboratory Values
Description: High density lipoprotein: males low 40 milligram/deciliter (mg/dL), high 80 mg/dL; females low 40 mg/dL, high 90 mg/dL. Low density lipoprotein (LDL): males and females low 70 mg/dL, high 139 mg/dL. Hemoglobin A1C (HBA1C): males and females low 4.3%, high 5.8%.
Time Frame: baseline through 18 weeks
Population: Analyzed were all participants who had baseline and post-baseline measurements. Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Number analyzed (Participants) | 100 | 39
participants
  Low high density lipoprotein (HDL); n=93, n=36 | 10 | 3
  High high density lipoprotein (HDL); n=95, n=37 | 5 | 1
  Low low density lipoprotein (LDL); n=97; n=37 | 1 | 1
  High low density lipoprotein (LDL); n=71, n=31 | 24 | 11
  Low hemoglobin A1C (HBA1C); n=100, n=39 | 1 | 1
  High hemoglobin A1C (HBA1C); n=97, n=38 | 2 | 0

ADVERSE EVENTS:
Arm/Group | Olanzapine Monotherapy | Olanzapine + Mood Stabilizer
Serious Adverse Events (participants affected / at risk) | 1/100 | 0/39
Other Adverse Events (participants affected / at risk) | 59/100 | 31/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine Monotherapy (N=100) | Olanzapine + Mood Stabilizer (N=39)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine Monotherapy (N=100) | Olanzapine + Mood Stabilizer (N=39)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Thirst (General disorders) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 17 (19) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (3)
Blood cholesterol increased (Investigations) | 3 (3) | 3 (3)
Blood triglycerides increased (Investigations) | 5 (5) | 6 (6)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2)
Low density lipoprotein increased (Investigations) | 1 (1) | 2 (2)
Weight increased (Investigations) | 9 (9) | 5 (5)
Somnolence (Nervous system disorders) | 15 (15) | 7 (8)
Depressive symptom (Psychiatric disorders) | 7 (7) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Identified errors were corrected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days